CLINICAL TRIAL: NCT01967472
Title: Adherence to Artemisinin-Based Combination Therapy (ACT) for the Treatment of Malaria in Sierra Leone
Brief Title: Adherence to Antimalarial Drugs in Sierra Leone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Malaria Control Program, Ministry of Health and Sanitation (Unknown); Pharmacy Board of Sierra Leone, Ministry of Health and Sanitation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-ACT-01
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- co-formulated Amodiaquine-Artesunate (Active Comparator): Sanofi Coarsucam Infant dose (2-12 months/4.5-8kg), amodiaquine:67.5mg/artesunate 25mg; 1 tablet once a day for 3 days.
  Sanofi Coarsucam Young Child (13-59 months/9-17kg), amodiaquine: 136mg/artesunate 50mg; 1 tablet once a day for 3 days.
  Interventions: Drug: amodiaquine-artesunate (AQAS) fixed-dose
- artemether-lumefantrine (Active Comparator): Novartis coartem infant dose (2-11 months/5-14kg), artemether 20mg/lumefantrine 120mg; 1 tablet twice a day for 3 days.
  Novartis coartem child dose (12-59 months/15-24kg), artemether 20mg/lumefantrine 120mg; 2 tablets twice a day for 3 days
  Interventions: Drug: Artemether-lumefantrine combination (AL) dispersable

INTERVENTIONS:
Drug: amodiaquine-artesunate (AQAS) fixed-dose
  Other Names: coarsucam, winthrop, co-formulated
  Arms: co-formulated Amodiaquine-Artesunate
Drug: Artemether-lumefantrine combination (AL) dispersable
  Other Names: coartem, AL, locally all Artemether-lumefantrine called 'lokmal'
  Arms: artemether-lumefantrine

SUMMARY:
The aim of this study is to address this gap in knowledge by measuring the level of patient adherence to co-formulated amodiaquine and artesunate (AQ-AS) compared to artemether-lumefantrine (AL) under routine conditions in Sierra Leone and explore the key factors that influence adherence. This will be addressed through a mixed methods study that will provide not only a measurement of adherence ACTs and malaria test results, but will also provide contextual information in order to better understand factors that affect adherence. Data will be collected through a series of interviews with health workers and parents/caregivers and through observations of patient-provider consultations.

The first stage of the study begins with semi-structured interviews and observations of patients/caretakers' consultations with health workers and will look at how health workers diagnose and treat malaria. This will be followed by short exit interviews at the health facility with caregivers to assess patient satisfaction with services, as well as to test the consistency between the data obtained through structured observations and the exit interviews.

Follow-up surveys at the homes of patients will be used to measure and compare the adherence of participants to two different ACTs (AQAS and AL) formulations and potential factors that affect adherence. Additionally, data will be collected using in-depth interviews to collect supplementary information in order to discover, in more detail, factors that may affect behavioral choices and/or attitudes with regard to adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a child between 6 to 59 months
* Visiting health facility for treatment of fever
* Do not have signs of severe disease
* Are not being referred to another health facility
* Living within a defined distance from the health facility (<8 km/ 5 miles)
* Have not taken part in the study already or are not part of a household that has already taken part in the study
* Responsible caretakers/parents provide additional informed consent

Exclusion Criteria:

-

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1145 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Adherence | Day 4
  Adherence is measured on the day following the last day of treatment. Adherence is defined as taking all of the prescribed dose at the correct time.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Banek, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Sierra Leone (2):
  - George Brook Health Center, Freetown
  - Ross Road Health Facility, Freetown

REFERENCES:
- [Derived] Banek K, Webb EL, Smith SJ, Chandramohan D, Staedke SG. Adherence to treatment with artemether-lumefantrine or amodiaquine-artesunate for uncomplicated malaria in children in Sierra Leone: a randomized trial. Malar J. 2018 Jun 4;17(1):222. doi: 10.1186/s12936-018-2370-x. PMID 29866192